CLINICAL TRIAL: NCT03011047
Title: Efficacy of Endoscopic Transantral Versus Transorbital Surgical Approaches in the Repair of Orbital Blow-Out Fractures-Randomized Clinical Trial.
Brief Title: Efficacy of Endoscopic Transantral Surgical Approach in the Repair of Orbital Blow-Out Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nahla Mahmoud Awad (Other)
Responsible Party: Sponsor-Investigator, Nahla Mahmoud Awad, Assistant lecturer , Oral and Maxillofacial surgery Department, Faculty of Oral & Dental Medicine Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-1-1
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Orbital Floor Fracture
Keywords: endoscopic, trans-antral, subciliary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic trans-antral approach (Experimental): The maxillary sinus and prolapsed orbital contents will be visualized employing a 30-degree endoscope for the repair of orbital blow out fracture (sinus scope 4 mm, 30 degrees short one 17 cm).
  Interventions: Procedure: endoscopic trans-antral approach
- trans-orbital surgical approach (Active Comparator): trans-orbital surgical approach through the lower eyelid Sub-ciliary incision ( through the lower eyelid) The skin incision is made just below the eyelashes.
  Interventions: Procedure: trans-orbital surgical approach

INTERVENTIONS:
Procedure: endoscopic trans-antral approach — new surgical approach to repair the orbital floor fractures through the maxillary sinus
  Other Names: trans-maxillary
  Arms: endoscopic trans-antral approach
Procedure: trans-orbital surgical approach — through the lower eyelid below the eyelashes ,then down to bone the herniated orbital content will be reduced through this incision traditional surgical approach to repair orbital floor fractures
  Other Names: sub-ciliary incision; lower eyelid incision; skin incision
  Arms: trans-orbital surgical approach

SUMMARY:
Aim of this study is to assess the efficacy of endoscopic trans-maxillary surgical approach versus traditional trans-orbital surgical approach (control group) in orbital blow out fractures in terms of postoperative clinical and digital radio-graphical assessments.

DETAILED DESCRIPTION:
(N.M) Operator, data entry & corresponding author; Assistant lecturer , surgery department .

(I.E) Main supervisor, data monitoring & auditing; Professor, surgery department.

(R.H) Co-supervisor, data entry & auditing; Lecturer, surgery department . (AM) Assistant lecturer, surgery department .Faculty of Oral & Dental Medicine Cairo University outcome assessors and data collection.

(YA) Assistant Lecturer of Surgery department , faculty of oral and dental medicine - Cairo University , for baseline data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants consents.

intervention:

Preoperative preparation:

Preoperative cone beam CT. A clearance from the ophthalmology department after examination of papillary reflexes, motility restriction and measurement of the visual acuity.

Laboratory Investigations: blood picture, liver functions, kidneys functions,coagulation profile Informed consent signed by the patient. (NM and RH) will perform all procedures under general anesthesia . Intervention :Endoscopic trans-maxillary (through the maxillary sinus) surgical approach.

control group: Traditional trans-orbital surgical approaches. follow up clinically and radio-graphically for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral/bilateral orbital blow out fractures.
2. Positive forced-duction test. ( to ensure the muscular entrapment).

Exclusion Criteria:

1. Medical condition affecting bone healing.
2. Medically compromised conditions, not proper candidate for general anesthesia.
3. Tumor case encroaching on the orbital floor.
4. Pathological orbital blow out fractures.
5. Allergy/ metal hypersensitivity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2017-08-18 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Diplopia resolution using Forced duction test positive/negative | 6 months
  subjective patient assessment

SECONDARY OUTCOMES:
Fracture reduction Digital radiography (Cone beam CT) | 6 months
Enophthalmus correction. Digital radiography (Cone beam CT) | 6 months
  mm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed elkhadem, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided